CLINICAL TRIAL: NCT07223385
Title: High Cardiovascular Risk Intervention With Cardio-Oncology Consultation for Prostate Cancer Following Androgen Receptor Pathway Inhibitor (ARPI) Therapy (Heart-Safe)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Katelyn Atkins, Sponsor-Investigator, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IIT2025-09-BALLAS-ATKINS-HEART
Record Dates: First submitted 2025-10-29; First posted 2025-10-31 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer (Diagnosis); Prostate Cancer Stage IV; CV Risk
Keywords: High-Risk; Lymph-node positive; ARPI Therapy; CV Risk Factors
MeSH Terms: conditions — Prostatic Neoplasms; Disease

STUDY DESIGN:
Intervention Model Description: Following eligibility verification, randomization will occur in REDCap via the Randomization Module. Patients will be randomized in a 1:1 ratio to (A) cardio-oncology management guidelines-based care vs. (B) notification to their primary care physician and/or general cardiologist of ARPI therapy initiation and recommendation for CV risk optimization (control) using stratified block randomization. Refer to section 10.0 for stratification methodology.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardo-Oncolody Referral (Experimental): Referral to cardio-oncology for guidelines-based personalized cardio-oncology management
  Interventions: Other: Cardio-Oncology Referral
- PCP/General Cardiology Care (Active Comparator): Notification to patient's primary care physician and/or general cardiologist and recommendation for CV risk optimization after initiation of ARPI therapy
  Interventions: Other: Notification to PCP/General Cardiologist

INTERVENTIONS:
Other: Cardio-Oncology Referral — Referral to cardio-oncology for guidelines-based personalized cardio-oncology management
  Arms: Cardo-Oncolody Referral
Other: Notification to PCP/General Cardiologist — Notification to patient's primary care physician and/or general cardiologist and recommendation for CV risk optimization after initiation of ARPI therapy
  Arms: PCP/General Cardiology Care

SUMMARY:
In patients with prostate cancer (PC), cardiovascular disease (CVD) causes significant morbidity and is the second leading cause of death. Both pre-existing CVD and the use of androgen deprivation therapy (ADT)-a key cornerstone of treatment for men with locally advanced or metastatic PC1,2 contribute to increased CV risk. ADT has been associated with adverse metabolic effects, including increased central adiposity, elevated low-density lipoprotein (LDL) levels, impaired glycemic control, and arterial wall remodeling and endothelial dysfunction

The data demonstrates that for most patients, the status quo is insufficient6 and there remains a critical gap in the early identification of high CV-risk PC patients who may benefit most from aggressive risk mitigation strategies. Mitigation strategies, like the addition of statins as primary prevention, have shown decrease in MI/CHD death across thousands of patients. Age-related expansion of hematopoietic clones carrying recurrent somatic mutations, termed clonal hematopoiesis of indeterminate potential (CHIP) has recently been identified as a significant driver of atherosclerosis, doubling the risk of coronary heart disease. Notably, while CHIP is detectable in ~10% of persons over 70 years old, it is enriched in patients with solid malignancies, and radiotherapy exposure is among the most decisive risk factors for developing CHIP12-15. The inflammation-related metabolic signals are activated androgen signaling and exacerbated in patients with CHIP. However, the mechanistic link and clinical consequence are less understood. Therefore, it is critical to study the CV impact of CHIP and metabolic perturbations in patients with PC treated with ARSI therapy.

We plan to address these critical gaps by testing our innovative hypothesis that early cardio-oncology intervention with aggressive guidelines-based CV optimization during ARPI therapy will reduce CV risk and that CHIP and metabolomics will help identify adverse metabolic remodeling to improve CV risk prediction.

Robust epidemiological and clinical trial data consistently demonstrate that patients with PC are poorly optimized from a CV risk modification perspective, and existing CV risk models do not perform well in patients with cancer. The data demonstrates that for most patients, the status quo is insufficient and there remains a critical gap in the early identification of high CV-risk PC patients who may benefit most from aggressive risk mitigation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer with localized, very-high risk, lymph-node positive, and/or metastatic (Stage IV) disease.
* Being treated with ARPI therapy with intended duration ≥ 18 months.
* Age > 65 years old and at least one CV risk factor, or age 45-65 years with at least two CV risk factors:

  * Hypertension
  * Hyperlipidemia
  * Diabetes mellitus
  * Family history of early CAD (male first-degree relative (father or brother) with CAD before age 55; female first-degree relative (mother or sister) with CAD before age 65)
  * Presence of coronary artery calcium (CAC) on chest CT imaging
* ECOG 0-2
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Prior ARPI therapy exposure > 6 months duration.
* Established care with cardio-oncologist (cardiologist with expertise in CV risks of cancer and cardiotoxic cancer therapies).

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Rate of any CV medication Initiation and/or Change | 3 Months Post-Intervention
  To evaluate the rate of any CV medication initiation and/or change at 3-months following cardio-oncology consultation versus standard of care. Rate of any CV medication intervention at 3-months (Note: CV medication defined as: lipid-lowering, anti-hypertensive, anti-anginal, anti-platelet, anti-arrhythmic, heart failure medications)

SECONDARY OUTCOMES:
The Rate of Compliance with CV Therapeutic Medication Intervention | 6 and 12 Months Post Intervention
  To determine the rate of compliance with CV therapeutic medication intervention at 6 and 12 months
Rate of Statin Intervetion | 3 Months Post Intervention
  To determine the rate of statin intervention at 3 months
Rate of Compliance with Statin Medication Intervention | 6 and 12 Months Post Intervention
  To determine the rate of compliance with statin medication intervention at 6 and 12 months
Rate of any CV Medication Intervention | 6 Months Post-Intervention
  To determine the rate of any CV medication intervention at 6 months
Changes in Biological CV Risk Factor | 3, 6, and 12 Month Post-Intervention
  To assess changes in biological CV risk factors (low density lipoprotein [LDL])
Changes in Biological CV Risk Factor | 3, 6, and 12 Month Post-Intervention
  To assess changes in biological CV risk factors (systolic blood pressure)
Changes in Biological CV Risk Factor | 3, 6, and 12 Month Post-Intervention
  To assess changes in biological CV risk factors (hemoglobin A1c)
Changes in Biological CV Risk Factor | 3, 6, and 12 Month Post-Intervention
  To assess changes in biological CV risk factors (body mass index)
Rate of Coronary Artery Disease Testing | 3, 6, and 12 Month Post-Intervention
  To determine the rate of coronary artery disease (CAD) testing (coronary CT angiograms, CAC scans, stress tests, and invasive coronary angiograms)
Rate of new CV or Cardiac Diagnosis | 3, 6, and 12 Month Post-Intervention
  To determine the rate of new CV or cardiac diagnosis
One-Year MACE Rate | 12 Months Post-Intervention
  To determine the one-year MACE rate
Rate of Grade ≥ 2 Cardiac CTCAE | 12 Month Post-Intervention
  To determine one-year rate of grade ≥ 2 cardiac common terminology criteria for adverse events (CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Katelyn Atkins, MD, PhD, Principal Investigator — Cedars-Sinai Medical Center; Leslie Ballas, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No